CLINICAL TRIAL: NCT04080141
Title: Therapeutic Termination of Pregnancy: Maternal and Paternal Mental Health Before and in the Long-term
Brief Title: Therapeutic Termination of Pregnancy and Psychiatric Implications
Acronym: TTOP_PSY
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: 981/b
Record Dates: First submitted 2019-07-26; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Therapeutic Abortion With Complications; Personality Disorders; Trauma, Psychological; Reproductive Behavior; Post Traumatic Stress Disorder; Depression, Reactive
Keywords: Therapeutic Abortion; Personality Disorders; Childhood Trauma; Post Traumatic Stress Disorder; Depression
MeSH Terms: conditions — Personality Disorders; Psychological Trauma; Reproductive Behavior; Stress Disorders, Post-Traumatic; Adjustment Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD+: Subjects with personality disorder
  Interventions: Diagnostic Test: Multiple psychometric questionnaire; Procedure: Clinical psychiatric examination
- PD-: Subjects without personality disorder
  Interventions: Diagnostic Test: Multiple psychometric questionnaire; Procedure: Clinical psychiatric examination

INTERVENTIONS:
Diagnostic Test: Multiple psychometric questionnaire — At the time of first contact (T0) only women were subjected to Hamilton's rating scale for depression (HRSD or HAM-D), Hamilton's rating scale for anxiety (HRSA or HAM-A), Beck Depression Inventory (BDI-II). At the follow up after 1 year from the first examination (T1) they were subjected to a questionnaire with multiple psychometric tests for mother and her partner. The female version included Post-traumatic stress disorder checklist (PCL-5), Iowa Personality Disorder Screen (IPDS), Beck Depression Inventory (BDI-II), Connor-Davidson Resilience Scale 10 (CD-RISC 10) and Short-Form Questionnaire on childhood trauma (CTQ-SF). The male version included Post-traumatic stress disorder checklist (PCL-5), Iowa Personality Disorder Screen (IPDS), Connor-Davidson Resilience Scale 10 (CD-RISC 10) and Short-Form Questionnaire on childhood trauma (CTQ-SF).
Procedure: Clinical psychiatric examination — At the time of first contact (T0) only women were subjected to psychiatric clinical examination

SUMMARY:
25 parental couples, with a prenatal diagnosis of fetal abnormality, had psychiatric evaluation for eligibility before TToP and after one year from the procedure. Women and unborn's fathers were also subjected to different psychometric questionnaires (HAM-D, HAM-A, BDI-II, PCL-5, IPDS, CTQ, CD-RISC-10).

DETAILED DESCRIPTION:
The therapeutic interruption of pregnancy (TTOP) may have psychiatric outcomes like depression, anxiety and post-traumatic stress disorder (PTSD). Personality issues, childhood traumas and paternal consequences are too little investigated in current Literature.

The investigator's aim is exploring the contribution of maternal personality disorders and maternal history of childhood traumas to psychiatric outcomes after a TToP, paternal psychiatric outcomes and their role on their partner's psychopathological and psychiatric outcomes.

25 couples, with a prenatal diagnosis of fetal abnormality, had psychiatric evaluation for eligibility before TToP and after one year from the procedure. Women and unborn's fathers were also subjected to different psychometric questionnaires (HAM-D, HAM-A, BDI-II, PCL-5, IPDS, CTQ, CD-RISC-10).

At the time of first contact (T0) only women were subjected to a psychiatric clinical examination in order to evaluate their legal eligibility to TToP, according to Italian Law n. 194/78. At T0 women were also subjected to Hamilton's rating scale for depression (HRSD or HAM-D), Hamilton's rating scale for anxiety (HRSA or HAM-A), Beck Depression Inventory (BDI-II). At the follow up after 1 year from the first examination (T1) the parental couples were subjected to a questionnaire with multiple psychometric tests for mother and her partner. The female version included Post-traumatic stress disorder checklist (PCL-5), Iowa Personality Disorder Screen (IPDS), Beck Depression Inventory (BDI-II), Connor-Davidson Resilience Scale 10 (CD-RISC 10) and Short-Form Questionnaire on childhood trauma (CTQ-SF). The male version included Post-traumatic stress disorder checklist (PCL-5), Iowa Personality Disorder Screen (IPDS), Connor-Davidson Resilience Scale 10 (CD-RISC 10) and Short-Form Questionnaire on childhood trauma (CTQ-SF).

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Prenatal diagnosis of fetal abnormality
* Adequate comprehension
* Legal eligibility to TToP procedure after psychiatric clinical evaluation
* Acceptance on a voluntary basis

Exclusion Criteria:

* Incapacity
* Acute psychosis

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 45 parental couples (90 subjects: 45 women and 45 men) with a prenatal diagnosis of fetral abnormality followed by Obstetrical Department of ASST Monza
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms in women | 1 year
  Change from Baseline in number of women with depressive symptoms at 1 year after TToP assessed with the Beck Depression Inventory, which measure the severity of depressive symptoms. The long form of the Beck Depression Inventory is composed of 21 questions or items, each with four possible responses. Each response is assigned a score ranging from zero to three, indicating the severity of the symptom. The sum of all item scores indicates the severity of depression. Scores from 0 to 9 represent minimal depressive symptoms, scores of 10 to 16 indicate mild depression, scores of 17 to 29 indicate moderate depression, and scores of 30 to 63 indicate severe depression. So, a higher value at the Beck Depression Inventory represent a worse outcome.
Post-traumatic stress disorder in women | 1 year
  Change from Baseline in number of women with post-traumatic symptoms at 1 year after TToP assessed with the PTSD Checklist 5, which is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. Items are summed to provide a total score. PCL-5 cut-point of 33 appears to be a reasonable value to use for provisional PTSD diagnosis. Severity can be determined adding scores of each item together to determine a total score. The range is 0-80 and a higher value represent a worse outcome

SECONDARY OUTCOMES:
Depressive symptoms after TToP in men | 1 year
  Change from Baseline in number of men with depressive symptoms at 1 year after TToP assessed with the Beck Depression Inventory, which measure the severity of depressive symptoms. The long form of the Beck Depression Inventory is composed of 21 questions or items, each with four possible responses. Each response is assigned a score ranging from zero to three, indicating the severity of the symptom. The sum of all item scores indicates the severity of depression. Scores from 0 to 9 represent minimal depressive symptoms, scores of 10 to 16 indicate mild depression, scores of 17 to 29 indicate moderate depression, and scores of 30 to 63 indicate severe depression. So, a higher value at the Beck Depression Inventory represent a worse outcome.
Post-traumatic stress disorder after TToP in men | 1 year
  Change from Baseline in number of men with post-traumatic symptoms at 1 year after TToP assessed with the PTSD Checklist 5 (PCL-5), which is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. Items are summed to provide a total score. PCL-5 cut-point of 33 appears to be a reasonable value to use for provisional PTSD diagnosis. Severity can be determined adding scores of each item together to determine a total score. The range is 0-80 and a higher value represent a worse outcome
Participants with personality disorder | 1 year
  Number of participants with personality disorder assessed with the Iowa Personality Disorder Screen, which is a 11-item screening instrument used to evaluate the presence of a personality disorder. Each item is scored dichotomously by Yes/No, giving individual IPDS scores ranging from 0 to 11. A cut off>4 positive items indicates the presence of a personality disorder. A higher value represent a worse outcome
Participants with childhood trauma | 1 year
  Number of participants with a childhood trauma assessed with the Childhood Trauma Questionnaire, which is a standardized, retrospective 28-item self-report inventory that measures the severity of different types of childhood trauma, producing five clinical subscales each comprised of five items: Emotional Abuse, Physical Abuse, Sexual Abuse, Emotional Neglect, Physical Neglect. Participants respond to each item in the context of "when you were growing up" and answer according to a five-point Likert scale ranging from "never" = 1 to "very often" = 5, producing scores of 5 to 25 for each trauma subscale. A cut off>5 points in every subscale indicates the presence of that particular traumatic experience. A higher score in every subscale represent a worse outcome and a more severe type of childhood trauma
Role of personality disorders on depressive symptoms after TToP | 1 year
  Difference in number of patients with depressive symptoms assessed with the Beck Depression Inventory (BDI, previously described) between participants with a personality disorder (PD+ group) and participants without a personality disorder (PD- group). This difference will be assessed with a statistical analysis. A higher number of patients with depressive symptoms in one of the two groups represent a worse outcome in that group
Role of personality disorders on post-traumatic symptoms after TToP | 1 year
  Difference in number of patients with post-traumatic symptoms assessed with the PTSD Checklist 5 (PCL-5, previously described) between participants with a personality disorder (PD+ group) and participants without a personality disorder (PD- group). This difference will be assessed with a statistical analysis. A higher number of patients with post-traumatic symptoms in one of the two groups represent a worse outcome in that group

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rasch V, Gammeltoft T, Knudsen LB, Tobiassen C, Ginzel A, Kempf L. Induced abortion in Denmark: effect of socio-economic situation and country of birth. Eur J Public Health. 2008 Apr;18(2):144-9. doi: 10.1093/eurpub/ckm112. Epub 2007 Dec 7. PMID 18065434
- [Background] Uria M, Mosquera C. Legal abortion in Asturias (Spain) after the 1985 law: sociodemographic characteristics of women applying for abortion. Eur J Epidemiol. 1999 Jan;15(1):59-64. doi: 10.1023/a:1007541904470. PMID 10098997
- [Background] Dehlendorf C, Harris LH, Weitz TA. Disparities in abortion rates: a public health approach. Am J Public Health. 2013 Oct;103(10):1772-9. doi: 10.2105/AJPH.2013.301339. Epub 2013 Aug 15. PMID 23948010
- [Background] Taft AJ, Watson LF. Termination of pregnancy: associations with partner violence and other factors in a national cohort of young Australian women. Aust N Z J Public Health. 2007 Apr;31(2):135-42. doi: 10.1111/j.1753-6405.2007.00031.x. PMID 17461004
- [Background] Dehlendorf C, Weitz T. Access to abortion services: a neglected health disparity. J Health Care Poor Underserved. 2011 May;22(2):415-21. doi: 10.1353/hpu.2011.0064. PMID 21551921
- [Background] Perez G, Ruiz-Munoz D, Gotsens M, Cases MC, Rodriguez-Sanz M. Social and economic inequalities in induced abortion in Spain as a function of individual and contextual factors. Eur J Public Health. 2014 Feb;24(1):162-9. doi: 10.1093/eurpub/ckt104. Epub 2013 Jul 31. PMID 23902666
- [Background] Taft AJ, Watson LF, Lee C. Violence against young Australian women and association with reproductive events: a cross-sectional analysis of a national population sample. Aust N Z J Public Health. 2004 Aug;28(4):324-9. doi: 10.1111/j.1467-842x.2004.tb00438.x. PMID 15704695
- [Background] Major B, Appelbaum M, Beckman L, Dutton MA, Russo NF, West C. Abortion and mental health: Evaluating the evidence. Am Psychol. 2009 Dec;64(9):863-90. doi: 10.1037/a0017497. PMID 19968372
- [Background] Steinberg JR, Finer LB. Examining the association of abortion history and current mental health: A reanalysis of the National Comorbidity Survey using a common-risk-factors model. Soc Sci Med. 2011 Jan;72(1):72-82. doi: 10.1016/j.socscimed.2010.10.006. Epub 2010 Oct 23. PMID 21122964
- [Background] Mota NP, Burnett M, Sareen J. Associations between abortion, mental disorders, and suicidal behaviour in a nationally representative sample. Can J Psychiatry. 2010 Apr;55(4):239-47. doi: 10.1177/070674371005500407. PMID 20416147
- [Background] Munk-Olsen T, Laursen TM, Pedersen CB, Lidegaard O, Mortensen PB. First-time first-trimester induced abortion and risk of readmission to a psychiatric hospital in women with a history of treated mental disorder. Arch Gen Psychiatry. 2012 Feb;69(2):159-65. doi: 10.1001/archgenpsychiatry.2011.153. PMID 22310504
- [Background] van Ditzhuijzen J, ten Have M, de Graaf R, van Nijnatten CH, Vollebergh WA. Psychiatric history of women who have had an abortion. J Psychiatr Res. 2013 Nov;47(11):1737-43. doi: 10.1016/j.jpsychires.2013.07.024. Epub 2013 Aug 12. PMID 23941742
- [Background] Wallin Lundell I, Sundstrom Poromaa I, Frans O, Helstrom L, Hogberg U, Moby L, Nyberg S, Sydsjo G, Georgsson Ohman S, Ostlund I, Skoog Svanberg A. The prevalence of posttraumatic stress among women requesting induced abortion. Eur J Contracept Reprod Health Care. 2013 Dec;18(6):480-8. doi: 10.3109/13625187.2013.828030. Epub 2013 Aug 26. PMID 23978220
- [Background] Simoila L, Isometsa E, Gissler M, Suvisaari J, Sailas E, Halmesmaki E, Lindberg N. Schizophrenia and induced abortions: A national register-based follow-up study among Finnish women born between 1965-1980 with schizophrenia or schizoaffective disorder. Schizophr Res. 2018 Feb;192:142-147. doi: 10.1016/j.schres.2017.05.039. Epub 2017 Jun 12. PMID 28615119
- [Background] O'Brien KM, Whelan DR, Sandler DP, Hall JE, Weinberg CR. Predictors and long-term health outcomes of eating disorders. PLoS One. 2017 Jul 10;12(7):e0181104. doi: 10.1371/journal.pone.0181104. eCollection 2017. PMID 28700663
- [Background] Roller CG. Sexually compulsive/addictive behaviors in women: a women's healthcare issue. J Midwifery Womens Health. 2007 Sep-Oct;52(5):486-91. doi: 10.1016/j.jmwh.2007.03.014. PMID 17826712
- [Background] De Genna NM, Feske U, Larkby C, Angiolieri T, Gold MA. Pregnancies, abortions, and births among women with and without borderline personality disorder. Womens Health Issues. 2012 Jul-Aug;22(4):e371-7. doi: 10.1016/j.whi.2012.05.002. PMID 22749198
- [Background] Bleil ME, Adler NE, Pasch LA, Sternfeld B, Reijo-Pera RA, Cedars MI. Adverse childhood experiences and repeat induced abortion. Am J Obstet Gynecol. 2011 Feb;204(2):122.e1-6. doi: 10.1016/j.ajog.2010.09.029. Epub 2010 Nov 11. PMID 21074137
- [Background] Niswander KR, Singer J, Singer M. Psychological reaction to therapeutic abortion. II. Objective response. Am J Obstet Gynecol. 1972 Sep 1;114(1):29-33. doi: 10.1016/0002-9378(72)90284-0. No abstract available. PMID 4404655
- [Background] Cohen L, Roth S. Coping with abortion. J Human Stress. 1984 Fall;10(3):140-5. doi: 10.1080/0097840X.1984.9934968. PMID 6520395
- [Background] Freeman EW, Rickels K, Huggins GR, Garcia CR, Polin J. Emotional distress patterns among women having first or repeat abortions. Obstet Gynecol. 1980 May;55(5):630-6. PMID 7366922
- [Background] Zolese G, Blacker CV. The psychological complications of therapeutic abortion. Br J Psychiatry. 1992 Jun;160:742-9. doi: 10.1192/bjp.160.6.742. PMID 1617354
- [Background] Smith EM. A follow-up study of women who request abortion. Am J Orthopsychiatry. 1973 Jul;43(4):574-85. doi: 10.1111/j.1939-0025.1973.tb00826.x. No abstract available. PMID 4716675
- [Background] Sharma V, Sommerdyk C, Sharma S. Post-abortion mania. Arch Womens Ment Health. 2013 Apr;16(2):167-9. doi: 10.1007/s00737-013-0328-0. Epub 2013 Feb 5. PMID 23381493
- [Background] Mahe V, Dumaine A. Oestrogen withdrawal associated psychoses. Acta Psychiatr Scand. 2001 Nov;104(5):323-31. doi: 10.1034/j.1600-0447.2001.00288.x. PMID 11722312
- [Background] Drower SJ, Nash ES. Therapeutic abortion on psychiatric grounds. Part I. A local study. S Afr Med J. 1978 Oct 7;54(15):604-8. PMID 741260
- [Background] Kersting A, Kroker K, Steinhard J, Hoernig-Franz I, Wesselmann U, Luedorff K, Ohrmann P, Arolt V, Suslow T. Psychological impact on women after second and third trimester termination of pregnancy due to fetal anomalies versus women after preterm birth--a 14-month follow up study. Arch Womens Ment Health. 2009 Aug;12(4):193-201. doi: 10.1007/s00737-009-0063-8. Epub 2009 Mar 6. PMID 19266250